CLINICAL TRIAL: NCT04761341
Title: FLIO and the Influence of Oral Lutein Supplementation on Macular Pigment
Acronym: FLOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FLOS Study
Record Dates: First submitted 2020-11-24; First posted 2021-02-18 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AMD (Experimental)
  Interventions: Drug: NUTROF TOTAL
- healthy control (Active Comparator)
  Interventions: Drug: NUTROF TOTAL

INTERVENTIONS:
Drug: NUTROF TOTAL — 1 per day over a course of 3 months

SUMMARY:
To investigate the effects of lutein supplementation on macular pigment density using FLIO and MPOD measurements in patients with age-related macular degeneration and healthy subjects over a course of 6 months.

DETAILED DESCRIPTION:
The human macula is a small area of the retina responsible for central vision. The yellow macular pigment contains three carotenoids, lutein ((3R,3'R,6'R)-lutein), zeaxanthin ((3R,3'R)-zeaxanthin), and meso-zeaxanthin ((3R,3'S;meso)-zeaxanthin). The human body is unable to synthesize lutein and zeaxanthin, thus needs to be obtained from dietary sources such as green leafy vegetables and supplements. The function of the macular pigment is to act as a filter by absorbing blue light that may attenuate photochemical damage of the retina. Furthermore, it protects against light induced oxidative damage by functioning as an antioxidant; scavenging free radicals. A growing body of evidence has established a link between the concentrations of the macular pigment carotenoids, the macular pigment optical density (MPOD) levels, visual performance and the risk of macular degeneration.

The ability of the macular pigment to absorb or filter blue light can be measured as macular pigment optical density (MPOD), which is directly related to the quantity of lutein and zeaxanthin in the macula. Furthermore, preliminary data showed that macular pigment can be evaluated using Fluorescence lifetime imaging ophthalmoscopy (FLIO). In a previous study the investigators have shown that FLIO provides contrast for macular pigment in patients with AMD and healthy subjects.

The purpose of this study is to investigate the effects of oral lutein supplementation on macular pigment density using FLIO and MPOD measurements in healthy subjects and patients with age-related macular degeneration (AMD) over a course of 6 months. Furthermore, the investigators will assess whether compositional and functional alterations of the gut metagenome may be related to age-related macular degeneration, and the effects of lutein supplementation on the gut. In addition, to blood samples, stool samples will be analysed accordingly to the currently running study on "The role of the gut metagenome on the development of ophthalmic diseases" ClinicalTrials.gov Identifier: NCT02438111. Faecal analyses will provide insight to how oral lutein supplementation effects the gut microbiota and how it is influenced by serum lutein Levels.

Objective is to investigate the effects of lutein supplementation on macular pigment density using FLIO and MPOD measurements in patients with age-related macular degeneration and healthy subjects over a course of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be willing to give written informed consent
* Probands 18 years of age or greater
* Both eyes will be assessed in the study

Exclusion Criteria:

* Opacities of ocular media excluding detailed observation of the retina
* Gastrointestinal diseases that could cause disturbance of dietary absorption
* History of lutein supplementation
* Allergy to lutein and zeaxanthin
* Missing compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2019-10-22 (Actual)

PRIMARY OUTCOMES:
MPOD (macular pigment optical Density) | 6 Months
  Method to detect changes in macular pigment optic Density using dual wavelength autofluorescence
Fluorescence Lifetime Imaging Ophthalmoscopy (FLIO) | 6 Months
  Retinal Autofluorescence lifetimes
Macular pigment screener (MPS) II | 6 Months
  Screening Method to detect changes in macular pigment optic Density using heterochromatic flicker photometry

SECONDARY OUTCOMES:
Contrast sensitivity | 6 Months
  Using Pelli-Robson charts
Visual acuity | 6 Months
  Visual acuity using ETDRS charts
Serum Lutein concentration | 6 Months
Stool Analysis namely taxonomic and functional characterization of gut microbiota | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Martin Zinkernagel, MD, PHD, Study Chair — Department of Ophthalmology, Inselspital, Bern University Hostpital, University of Bern, Bern, Switzerland
Locations (1):
- Department of Ophthalmology, Inselspital, Bern University Hostpital, University of Bern, Bern, Switzerland, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jaggi D, Solberg Y, Dysli C, Lincke J, Habra O, Wyss A, Wolf S, Zinkernagel M. Fluorescence lifetime imaging ophthalmoscopy and the influence of oral lutein/zeaxanthin supplementation on macular pigment (FLOS) - A pilot study. Clin Nutr ESPEN. 2023 Aug;56:127-134. doi: 10.1016/j.clnesp.2023.05.009. Epub 2023 May 15. PMID 37344061